CLINICAL TRIAL: NCT03039699
Title: International Multicenter, Double-blind, Randomized, Parallel Group Placebo-Controlled Clinical Trial of Efficacy and Safety of Ergoferon in the Treatment of Viral Intestinal Infections in Children
Brief Title: Clinical Trial of Efficacy and Safety of Ergoferon in the Treatment of Viral Intestinal Infections in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-ER-008
Record Dates: First submitted 2016-12-28; First posted 2017-02-01 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-11

CONDITIONS: Viral Intestinal Infection
MeSH Terms: interventions — ergoferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergoferon (Experimental): Tablet for oral use. Dose per administration - 1 tablet per intake (outside a meal/feeding). Within the first 2 hours - 1 tablet every 30 minutes, followed by 3 more tablets at time intervals equally separated throughout the rest of the day; from day 2 to day 5 - 1 tablet 3 times daily.
  Interventions: Drug: Ergoferon
- Placebo (Placebo Comparator): Tablet for oral use. Dose per administration - 1 tablet per intake (outside a meal/feeding). Within the first 2 hours - 1 tablet every 30 minutes, followed by 3 more tablets at time intervals equally separated throughout the rest of the day; from day 2 to day 5 - 1 tablet 3 times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergoferon
  Arms: Ergoferon
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to obtain additional data on efficacy and safety of Ergoferon in the treatment of viral intestinal infections in inpatient children.

DETAILED DESCRIPTION:
Design: a multicenter, double-blind, placebo-controlled, randomized clinical trial in parallel groups.

This study will enroll subjects of both sexes aged from 6 months to 6 years who are admitted to hospital within 48 h of the onset of acute intestinal infection (AII), presumably of viral aetiology. Patients to be enrolled in the screening will be children with typical viral gastroenteritis/enteritis symptoms. The key symptom is decreased in the consistency of stools (loose or liquid) and increased in the frequency of its evacuations (at list 3 time daily). Virus detection in stool samples will be performed by polymerase chain reaction (PCR).

After the parent/adopter signs a parents/adopters information sheet (Informed Consent form) for the child's participation in the clinical trial, the recording of medical history data, a medical examination including the evaluation of symptoms on the Clinical Dehydration Scale (CDS) by pediatrician, and laboratory tests will be performed during Visit 1 (Day 1). If inclusion criteria are met and non-inclusion criteria are absent (day 1), the patient will be included in the trial and randomized to administer either Ergoferon or Placebo.

In addition to the standard/pathogenetic therapies, group 1 patients will take Ergoferon following a 5-day regimen, whereas group 2 patients will receive Placebo. The parents/adopters of the patient will be provided with a patient diary and instructed how to complete the diary.

Before treatment stool specimens will be collected from the patients for detection and differentiation of Rotavirus A, Norovirus 2 genotype, Astrovirus, Adenovirus F, Shigella spp., enteroinvasive E.coli (EIEC), Salmonella spp., and thermophilic Campylobacter spp. using a PCR assay to diagnose the etiology of intestinal infection. In total, the patients will be monitored for 10 days (screening, randomization, treatment initiation - Day 1; the treatment on Days 1-5; observation in hospital - Day 6, and follow-up period - Day 7-10). During the treatment and inpatient observation periods (Days 1-6, Visits 1-6), the patients will be examined daily by a pediatrician, and the examination results, including the CDS scores, will be recorded in source documents. The patient's parent/adopter will complete the patient diary every day, recording the presence/absence of diarrhea signs, vomiting, and body temperature. The pediatrician will check them each time for the correctness of completion. On day 10 (after hospital discharge), Visit 7 will be done (as an in-person visit (a hospital or calling a doctor) or a distance, 'phone' visit) to interview the parents/adopters about the patient's health, presence of any complications, and use of medications (the pediatrician will use this information to complete a questionnaire). Collection of stool specimens and repeat PCR for Rotaviruses/Noroviruses/Astroviruses/Adenoviruses, Shigella spp., EIEC, Salmonella spp., and Campylobacter spp. will be performed on Days 3, 4, and 6 of inpatient observation and after discharge from the hospital (Day 10); collection of blood and urine specimens for safety tests will be carried out at baseline and before hospital discharge (day 6). The recording of the intake of study therapies and of concomitant medications as well as the assessment of compliance with and safety of the study therapies will be performed on Days 2-6 and 10.

Patients who recovered while in hospital and are discharged from the unit earlier than at 5 days will undergo the procedures of Visit 6, including the collection of biological specimens for PCR (efficacy evaluation) and biochemistry, blood test and urinalysis (safety assessment). The parents/adopters will be given the blister pack with the remaining study drug so that the patient can continue the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both gender aged from 6 months to 6 years, who have been admitted to infectious diseases unit.
2. Diarrhea (watery diarrhea at least 3 times a day).
3. CDS score of ≥1.
4. The first 48 hours from the onset of the first diarrhea episode.
5. Start of study treatment (Ergoferon/Placebo) within 12 hours after the start of the standard hospital therapy.
6. Availability of a patient information sheet (Informed Consent form) signed by the patient's parents/adopters to confirm the child's participation in the clinical trial signed by one parent/adopter of the patient.

Exclusion Criteria:

1. Suspected bacterial intestinal infection.
2. Suspected infectious diseases affecting other organ systems (e.g. pneumonia, meningitis, sepsis, otitis media, urinary tract infection, etc.).
3. Severe intestinal infection.
4. Severe dehydration (CDS score ≥7).
5. Anuria (acute kidney injury).
6. Medical history or prior diagnosis of serious diseases, including primary/secondary immunodeficiency, oncological disease, diabetes mellitus, infantile cerebral palsy, mucoviscidosis/cystic fibrosis etc.
7. Exacerbation, or decompensation of chronic disease, including diseases of the digestive system that would affect the patient's ability to participate in the clinical trial.
8. Malabsorption syndrome, including congenital or acquired lactose intolerance/lactase deficiency or any other disaccharidase deficiency and galactosemia.
9. Allergy/ intolerance to any of the components of medications used in the treatment.
10. Course intake of medicines listed in the section "Prohibited concomitant treatment" for 2 weeks prior to the enrollment in the trial.
11. Participation in other clinical trials within 3 months prior to the enrollment in this study.
12. Patients whose parents/adopters, from the investigator's point of view, will fail to comply with the observation requirements of the trial or with the dosing regimen of the study drugs.
13. Patient's parents/adopters are related to the research staff of the clinical investigative site who are directly involved in the trial or are the immediate family member of the researcher. The immediate family members include husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
14. The patient's parent/adopter works for MATERIA MEDICA HOLDING (i.e., is the company's employee, temporary contract worker or appointed official responsible for carrying out the research) or the immediate relative.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (12):
  - State budgetary Health Care institution of the Arkhangelsk region "Arkhangelsk Regional Pediatric Clinical Hospital named after PG Vyzhletsova", Arkhangelsk
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University" of the Ministry of Healthcare of the Russian Federation, Kazan'
  - Federal Budget Institution of Science "Central Research Institute of Epidemiology" of The Federal Service on Customers' Rights Protection and Human Well-being Surveillance, Moscow
  - Pirogov Russian National Research Medical University, Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Orenburg State Medical University" of the Ministry of Healthcare of the Russian Federation, Orenburg
  - Municipal Budgetary Health Care Institution "Semashko City Hospital №1 Rostov-on-Don ", Rostov-on-Don
  - Federal State Budgetary Educational Institution of Higher Education "Saint Petersburg State Pediatric Medical University" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - Sailnt Petersburg State Budgetary Health Care Institution "City Child Hospital №22", Saint Petersburg
  - Federal State Institution "Scientific Research Institute of Children's Infections Federal Biomedical Agency", Saint Petersburg
  - The State Budget Educational institution of High Professional Training Smolensk State Medical University of Ministry of Health Care of the Russian Federation, Smolensk
  - Federal State Budgetary Educational Institution of Higher Education "Yaroslavl State Medical University" of the Ministry of Healthcare of the Russian Federation, Yaroslavl
  - Federal State Budgetary Institution of Higher Professional Education "Urals State Medical University" of the Ministry of Healthcare of the Russian Federation, Yekaterinburg
- Scientific Research Institute of Virology of Ministry of Health of Republic Uzbekistan, Tashkent, Uzbekistan

RESULTS

PARTICIPANT FLOW:
Groups:
- Ergoferon: Within the first 2 hours - 1 tablet every 30 minutes, followed by 3 more tablets at time intervals equally separated throughout the rest of the day; from day 2 to day 5 - 1 tablet 3 times daily.
  Ergoferon
- Placebo: Within the first 2 hours - 1 tablet every 30 minutes, followed by 3 more tablets at time intervals equally separated throughout the rest of the day; from day 2 to day 5 - 1 tablet 3 times daily.
  Placebo
Period: Overall Study
Arm/Group | Ergoferon | Placebo
Started | 127 | 132
Completed | 105 | 97
Not Completed | 22 | 35
Not completed — Incorrect inclusion | 5 | 4
Not completed — Lack of data to assess study endpoint | 5 | 3
Not completed — Bacterial infection | 12 | 28

BASELINE CHARACTERISTICS:
Groups:
- Ergoferon: 1 tablet 3 times a day
  Ergoferon
- Placebo: 1 tablet 3 times a day
  Placebo
- Total: Total of all reporting groups
Arm/Group | Ergoferon | Placebo | Total
Number analyzed (Participants) | 127 | 132 | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 127 | 132 | 259
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.3 (1.5) | 2.3 (1.4) | 2.3 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 63 | 113
  Male | 77 | 69 | 146
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Uzbekistan | 53 | 56 | 109
  Russia | 74 | 76 | 150

OUTCOME MEASURES:

1. Primary Outcome: Average Diarrhea Duration.
Description: Diarrhea duration is considered as the time between receiving the first dose of investigational medicine /placebo and the normal consistency of stool pattern (to the previous stool consistency before diarrhea), i.e.
  1. time to the first loose stool which is followed by two normal consistency stools over 24 h (infants may have three episodes of loose stool over a 24-hour period), or
  2. time to ≤3 episodes of stool occurring over 24 h, at least 2 of which are normal consistency stools, or
  3. time to the absence of stools for ≥12 h which is not followed by new episodes of diarrhea (total stool frequency over 24 h - less than 3 times).
Time Frame: On days 1-10 of observation period.
Population: 2 patients in Ergoferon group and 2 patients in Placebo group had no primary outcome data
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 103 | 95
hours | 43.4 [37.9 to 49] | 54.7 [49 to 60.5]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.004, t-test, 2 sided

2. Secondary Outcome: Percentage of Patients Without Diarrhea.
Description: Based on medical records.
Time Frame: 48, 72 and 96 hours of the treatment.
Population: 2 patients in Ergoferon group and 2 patients in Placebo group had no primary outcome data
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 103 | 95
Participants
  48 hours | 62 | 41
  72 hours | 86 | 66
  96 hours | 98 | 88
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; 48 hours timepoint comparison; Test type: Superiority; p = 0.0675, Fisher Exact — p-value adjusted for multiple comparisons using Holm method
Statistical Analysis 2: Comparison: Ergoferon vs Placebo; 72 hours timepoint comparison; Test type: Superiority; p = 0.0675, Fisher Exact — p-value adjusted for multiple comparisons using Holm method
Statistical Analysis 3: Comparison: Ergoferon vs Placebo; 96 hours timepoint comparison; Test type: Superiority; p = 0.5569, Fisher Exact — p-value adjusted for multiple comparisons using Holm method

3. Secondary Outcome: Percentage of Patients With Recovery.
Description: Based on medical records. Recovery criteria: absence of diarrhea, vomiting, symptoms of dehydration, and increased body temperature (based on daily examinations by pediatrician).
Time Frame: 48, 72 and 96 hours of the treatment.
Population: 2 patients in Ergoferon group and 2 patients in Placebo group had no primary outcome data
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 103 | 95
Participants
  48 hours | 66 | 46
  72 hours | 88 | 68
  96 hours | 100 | 88
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; 48 hours timepoint comparison; Test type: Superiority; p = 0.0696, Fisher Exact — p-value adjusted for multiple comparisons using Holm method
Statistical Analysis 2: Comparison: Ergoferon vs Placebo; 72 hours timepoint comparison; Test type: Superiority; p = 0.0696, Fisher Exact — p-value adjusted for multiple comparisons using Holm method
Statistical Analysis 3: Comparison: Ergoferon vs Placebo; 96 hours timepoint comparison; Test type: Superiority; p = 0.1998, Fisher Exact — p-value adjusted for multiple comparisons using Holm method

4. Secondary Outcome: Average Illness Duration.
Description: From the enrollment to the recovery. Recovery criteria: absence of diarrhea, vomiting, symptoms of dehydration, and increased body temperature (based on daily examinations by pediatrician).
Time Frame: On days 1-10 of observation period.
Population: 2 patients in Ergoferon group and 2 patients in Placebo group had no primary outcome data
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 103 | 95
hours | 40.8 [35.3 to 46.3] | 53.0 [47.2 to 58.9]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.0039, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Total Clinical Dehydration Scale Score.
Description: Based on medical records. Clinical Dehydration Scale score is more or equal 1. Note: minimum values - 0 points, maximum values - 8 points. Interpretation: 0 points - no dehydration, from 1 to 4 points - light dehydration, 5-8 points - average/severe dehydration.
Time Frame: 24, 48, and 72 hours of the treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 105 | 97
score on a scale
  24 hours | 1.5 [1.3 to 1.8] | 1.5 [1.2 to 1.7]
  48 hours | 0.3 [0.2 to 0.5] | 0.3 [0.1 to 0.4]
  72 hours | 0.1 [0 to 0.2] | 0.1 [0 to 0.1]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.89, Mixed Models Analysis — The p-value associated with "treatment*visit" interaction of total CDS score from 24 hours to 48 and 72 hours of treatment between Ergoferon and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

6. Secondary Outcome: Average Vomiting Duration (if Any).
Description: Based on medical records.
Time Frame: On days 1-10 of observation period.
Population: Vomiting occured in 64.8% patients of Ergoferon group and 71.1% patients of placebo group.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 68 | 69
hours | 44.6 [35.1 to 54.1] | 57.9 [48.4 to 67.5]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.0044, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percentage of Patients With Negative PCR Tests.
Description: Based on medical records.
Time Frame: On days 3, 4, 6 and 10 of observation period.
Population: PCR tests on days 4, 6 and 10 were run on less patients due to technical issues in laboratory
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 81 | 71
Participants
  Day 3 | 5 | 7
  Day 4: number analyzed (Participants) | 77 | 69
  Day 4 | 12 | 9
  Day 6: number analyzed (Participants) | 80 | 69
  Day 6 | 15 | 21
  Day 10: number analyzed (Participants) | 73 | 69
  Day 10 | 25 | 29
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Day 3 comparison; Test type: Superiority; p = 0.5488, Fisher Exact — nonadjusted p-value
Statistical Analysis 2: Comparison: Ergoferon vs Placebo; Day 4 comparison; Test type: Superiority; p = 0.8140, Fisher Exact — nonadjusted p-value
Statistical Analysis 3: Comparison: Ergoferon vs Placebo; Day 6 comparison; Test type: Superiority; p = 0.1248, Fisher Exact — nonadjusted p-value
Statistical Analysis 4: Comparison: Ergoferon vs Placebo; Day 10 comparison; Test type: Superiority; p = 0.3889, Fisher Exact — nonadjusted p-value

8. Secondary Outcome: Percentage of Patients With Worsening of Illness and/or Hospital-acquired Infection.
Description: Based on medical records. Worsening of illness: an increase in dehydration scores and worsening of non-specific symptoms, as evidenced by a decline in general appearance, increasing fatigue and drowsiness, refusal to eat and drink, severe tachycardia/bradycardia, unstable hemodynamics, tachypnea, hypo- or hyperventilation, circulation disorders, peripheral cyanosis, sunken eyes, severe dryness of skin and mucous/tongue, poor tissue turgor, absent tears, persistent vomiting, anuria/acute kidney injury, seizure/convulsions, and meningismus. Hospital-acquired infection: a viral or bacterial infection (intestinal, respiratory or urinary tract infection, etc.) occurring after at least 48 h of hospital stay and confirmed by laboratory tests.
Time Frame: On days 1-10 of observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 105 | 97
Participants | 4 | 7
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.3593, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were collected for 10 days of the therapy and follow-up periods.
Description: Adverse/Serious adverse events were collected in patients of the Safety population (n=259).
Arm/Group | Ergoferon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/132
Serious Adverse Events (participants affected / at risk) | 2/127 | 0/132
Other Adverse Events (participants affected / at risk) | 10/127 | 5/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoferon (N=127) | Placebo (N=132)
Acute respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Purine metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Functional stomach upset. Disoder of purine metabolism (acetone vomiting).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoferon (N=127) | Placebo (N=132)
Acute nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Acute otitis media (Infections and infestations) | 0 (0) | 1 (1) — Left-sided otitis media (acute, non-suppurative)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Leukocytes in urine (Renal and urinary disorders) | 0 (0) | 1 (1) — An increase in the number of leukocytes in the urine.
Candida Infection (Infections and infestations) | 1 (1) | 1 (1)
Increased levels of ALT (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Increased levels of AST (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Increase in the percentage of lymphocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Decrease in the percentage of neutrophils
Positive test result for staphylococcus (Infections and infestations) | 1 (1) | 0 (0) — Positive result of isolation and identification of staphylococcus. Discharge of staphylococcus from the nasopharynx.
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) — The presence of blood in the stool.
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Herpangina caused by Coxsackie virus (Infections and infestations) | 1 (1) | 0 (0) — Vesicular pharyngitis
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperphosphaturia (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03039699/Prot_SAP_000.pdf